CLINICAL TRIAL: NCT06282016
Title: Risk Factors for Neuroendocrine Neoplasms: a Case-control Study Based on a Record Linkage of Registry and Claims Data
Brief Title: Risk Factors for Neuroendocrine Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Bavarian Cancer Registry (Other Government)
Collaborators: Bavarian Association of Statutory Health Insurance Accredited Physicians (Unknown)
Responsible Party: Sponsor
Other Study IDs: BKR-2024-001
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Neoplasm of Lung; Neuroendocrine Neoplasm of Gastrointestinal Tract (Disorder)
Keywords: Neuroendocrine neoplasms; Colorectal cancer; Risk factors; Case-Control Study; Cancer Registry
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Case-Control Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a neuroendocrine neoplasm of the bronchopulmonary or gastroenteropancreatic system diagnosed between 2021 and 2023
  Interventions: Other: Case-control study (no intervention)
- Controls: Patients without a neuroendocrine neoplasm of the bronchopulmonary or gastroenteropancreatic system diagnosed between 2021 and 2023 (=no documented diagnosis of neuroendocrine neoplasm of the bronchopulmonary or gastroenteropancreatic system in the Bavarian Cancer Registry)
  Interventions: Other: Case-control study (no intervention)

INTERVENTIONS:
Other: Case-control study (no intervention) — Observation of risk factors in cases and controls

SUMMARY:
Recent studies show an increase in neuroendocrine neoplasms, especially for the digestive tract. Previous studies suggest various risk factors that were observed for various tumor sites, e.g. a family history of cancer, tobacco and alcohol consumption as well as metabolic disorders including diabetes and obesity. A risk factor that has been little studied to date is depressive disorders, which could increase the risk of neuroendocrine neoplasms either independently or through associated risk behaviors and/or antidepressant medication. The aim of this study is to identify risk factors for neuroendocrine neoplasms based on a case-control study in order to better understand the increase of neuroendocrine neoplasms in recent decades. The study is based on a record linkage of data from the Bavarian Cancer Registry and data from the Bavarian Association of Statutory Health Insurance Accredited Physicians. While the data from the Bavarian Cancer Registry enables the identification of neuroendocrine neoplasms on the basis of histopathological findings and thus is the basis for selecting cases, the claims data from the Bavarian Association of Statutory Health Insurance Accredited Physicians provides the source population as well data on diagnoses and thus enables the investigation of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a statutory health insurance (about 85% of the population) and at least one outpatient physician contact in Bavaria between 2021 and 2023
* Residence in Bavaria

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases are defined as all persons with a malignant neuroendocrine neoplasm of the bronchopulmonary or gastroenteropancreatic system diagnosed between 2021 and 2023. Controls are defined as noncases in the source population of cases, i.e. persons with a statutory health insurance and at least one outpatient physician contact in Bavaria between 2021 and 2023, whose residence was in Bavaria. Two controls will be sampled for each case.
Sampling Method: Probability Sample
Enrollment: 14250 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assured NEN diagnosis of the BPS | 2021-2023
  Neuroendocrine neoplasm of the bronchopulmonary system
Assured NEN diagnosis of the GEPS | 2021-2023
  Neuroendocrine neoplasm of the gastroenteropancreatic system

SECONDARY OUTCOMES:
Assured NET diagnosis of the BPS | 2021-2023
  Neuroendocrine tumour of the bronchopulmonary system
Assured NEC diagnosis of the BPS | 2021-2023
  Neuroendocrine carcinoma of the bronchopulmonary system
Assured NET diagnosis of the GEPS | 2021-2023
  Neuroendocrine tumour of the gastroenteropancreatic system
Assured NEC diagnosis of the GEPS | 2021-2023
  Neuroendocrine carcinoma of the gastroenteropancreatic system

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Müller-Nordhorn, Principal Investigator — Bavarian Cancer Registry, Bavarian Health and Food Safety Authority; Martin Tauscher, Principal Investigator — Bavarian Association of Statutory Health Insurance Accredited Physicians
Locations (1):
- Bavarian Cancer Registry, Bavarian Health and Food Safety Authority, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voigtlander S, Gerlach R, Grundmann N, Donnachie E, Berger U, Hakimhashemi A, Meyer M, Tauscher M, Muller-Nordhorn J. Risk factors for neuroendocrine neoplasms: protocol for a case-control study based on a record linkage of registry and claims data. BMJ Open. 2025 May 23;15(5):e096273. doi: 10.1136/bmjopen-2024-096273. PMID 40409959